CLINICAL TRIAL: NCT01177410
Title: A Phase II, Randomized, Placebo-controlled, Double-blind, Multicenter, 12 Week Study to Assess the Efficacy and Safety of Mesalamine Granules 750 mg and 1,500 mg Capsules Administered Once Daily in the Treatment of Irritable Bowel Syndrome With Diarrhea
Brief Title: Mesalamine Granules for Irritable Bowel Syndrome (IBS) With Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGIB2051
Record Dates: First submitted 2010-07-30; First posted 2010-08-09 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS; Diarrhea; IBS-D; Irritable Bowel Syndrome; Abdominal pain; Bloating
MeSH Terms: conditions — Diarrhea; Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Mesalamine Granules 750 mg (Experimental)
  Interventions: Drug: Mesalamine Granules 750 mg
- Mesalamine Granules 1500 mg (Experimental)
  Interventions: Drug: Mesalamine Granules 1500 mg

INTERVENTIONS:
Drug: Placebo — placebo capsules once daily for 12 weeks
  Arms: Placebo
Drug: Mesalamine Granules 750 mg — 750 mg mesalamine granules once daily for 12 weeks
  Arms: Mesalamine Granules 750 mg
Drug: Mesalamine Granules 1500 mg — 1500 mg mesalamine granules once daily for 12 weeks
  Arms: Mesalamine Granules 1500 mg

SUMMARY:
The purpose of this study is to determine the daily dose of mesalamine granules that will provide adequate relief from symptoms of IBS with diarrhea.

ELIGIBILITY:
Inclusion Criteria:

Male or non-pregnant, non-lactating female subjects Diagnosed with IBS confirmed by the Rome III criteria

Meet the following IBS symptom scores in all categories during the diary eligibility period:

* An average daily score of greater than or equal to 3 for abdominal pain
* An average daily score of greater than or equal to 3 for bloating
* An average daily score of 5 or greater for stool consistency using the Bristol Stool Scale
* Does not have adequate relief of IBS symptoms (weekly reported) over the past 7 days on the first day of screening and on the day of randomization

Exclusion Criteria:

* Present with hard or lumpy stools (Type 1 or Type 2) on the Bristol Stool form Scale during the diary eligibility period
* history of inflammatory bowel disease
* has Type 1 or 2 diabetes
* pregnant or lactating
* history of HIV or hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Sherwood, Arkansas
  - Anaheim, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Bristol, Connecticut
  - Boynton Beach, Florida
  - St. Petersburg, Florida
  - Macon, Georgia
  - Shreveport, Louisiana
  - Ann Arbor, Michigan
  - Wyoming, Michigan
  - Mexico, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Greensboro, North Carolina
  - Plano, Texas
  - Ogden, Utah
  - Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period: 09Aug2010 to 16Aug2011. 20 Study Sites; US Only. Study locations were a variety including: Gastrointestinal, Family Practice, Medical Centers and/or University setting
Pre-assignment Details: Failure to meet baseline IBS symptom scores (based on diary responses)
Groups:
- Mesalamine Granules 1500 mg: Mesalamine Granules 1500 mg : 1500 mg mesalamine granules once daily for 12 weeks
- Mesalamine Granules 750 mg: Mesalamine Granules 750 mg : 750 mg mesalamine granules once daily for 12 weeks
- Placebo: Placebo : placebo capsules once daily for 12 weeks
Period: Overall Study
Arm/Group | Mesalamine Granules 1500 mg | Mesalamine Granules 750 mg | Placebo
Started | 51 | 47 | 50
Completed | 50 | 40 | 45
Not Completed | 1 | 7 | 5
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesalamine Granules 1500 mg | Mesalamine Granules 750 mg | Placebo | Total
Number analyzed (Participants) | 51 | 47 | 50 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 48 | 41 | 48 | 137
  >=65 years | 2 | 6 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.17) | 44.4 (16) | 44.6 (12.04) | 43.8 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 30 | 92
  Male | 19 | 17 | 20 | 56
Region of Enrollment [Number; unit: participants]
  United States | 51 | 47 | 50 | 148

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Subjects Who Are Monthly Responders in Both Abdominal Pain and Stool Consistency for at Least 2 Months During the 3-month Treatment Period
Description: A weekly responder in abdominal pain is defined as a ≥30% improvement from baseline in the weekly average abdominal pain score on a 10-point scale (0=no pain - 10= worst possible pain). A weekly responder in stool consistency is defined as ≥50% reduction in the number of days in a week with stool consistency of Type 6 or 7 compared with baseline using the Bristol Stool Scale. Monthly responders are subjects who are weekly responders in both abdominal pain and stool consistency for at least two out of four weeks.
Time Frame: 3 months
Population: Intent to Treat Population included all randomized subjects who ingested at least one dose of study drug. Analysis of study data was based on observed cases, missing data remained missing.
Measure: Number; unit: participants
Arm/Group | Mesalamine Granules 1500 mg | Mesalamine Granules 750 mg | Placebo
Number analyzed (Participants) | 51 | 47 | 50
participants | 24 | 15 | 14
Statistical Analysis 1: Comparison: Mesalamine Granules 1500 mg vs Mesalamine Granules 750 mg; Test type: Superiority or Other; p = 0.0432, Regression, Logistic; Odds Ratio (OR) = 2.369, 95% CI 2-sided [1.027 to 5.467]
Statistical Analysis 2: Comparison: Mesalamine Granules 750 mg vs Placebo; Test type: Superiority or Other; p = 0.6059, Regression, Logistic; Odds Ratio (OR) = 1.267, 95% CI 2-sided [0.515 to 3.115]

2. Primary Outcome: The Number of Months That Subjects Are Monthly Responders in Both IBS-related Abdominal Pain AND Stool Consistency During the Entire Three Months.
Description: as for outcome 1
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mesalamine Granules 1500 mg | Mesalamine Granules 750 mg | Placebo
Number analyzed (Participants) | 51 | 47 | 50
participants
  0 month | 18 | 27 | 28
  1 month | 9 | 5 | 8
  2 months | 13 | 5 | 6
  3 months | 11 | 10 | 8
Statistical Analysis 1: Comparison: Mesalamine Granules 1500 mg vs Placebo; Proportional odds model was used to compare the number of months the subjects are responders; Test type: Superiority or Other; p = 0.0327, Proportional Odds Model; Odds Ratio (OR) = 2.232, 95% CI 2-sided [1.068 to 4.664]
Statistical Analysis 2: Comparison: Mesalamine Granules 750 mg vs Placebo; Test type: Superiority or Other; p = 0.7260, Proportional Odds Model; Odds Ratio (OR) = 1.148, 95% CI 2-sided [0.531 to 2.483]

ADVERSE EVENTS:
Time Frame: Study Duration; Reported adverse events (AEs) include AEs observed over the 48 weeks of treatment.
Description: SAEs will be followed for up to 30 days post treatment
Arm/Group | Mesalamine Granules 1500 mg | Mesalamine Granules 750 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/47 | 0/50
Other Adverse Events (participants affected / at risk) | 15/51 | 9/47 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamine Granules 1500 mg (N=51) | Mesalamine Granules 750 mg (N=47) | Placebo (N=50)
Incision Site Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamine Granules 1500 mg (N=51) | Mesalamine Granules 750 mg (N=47) | Placebo (N=50)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 3 (3) | 2 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR shall not publish the results of the Study conducted at the INSTITUTION, unless they (i) obtain the prior written consent of SALIX for the publication; or (ii) withhold any publication for a period of two (2) years following the Completion of the Study by all participating institutions and investigators